CLINICAL TRIAL: NCT03142529
Title: Clinical Observation of Therapeutic Effects on Traditional Chinese Medicine Colon Dialysis Treating Non-dialysis End-Stage Kidney Disease
Brief Title: Traditional Chinese Medicine (TCM) Colon Dialysis Treats Non-dialysis End-Stage Kidney Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pang Peng (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Pang Peng, Principal Investigator, Jinan University Guangzhou
Organization: Jinan University Guangzhou (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRF-CD2017
Record Dates: First submitted 2017-04-20; First posted 2017-05-05 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Chronic Kidney Failure; End-Stage Kidney Disease
Keywords: Non dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Therapy (No Intervention): This arm is an control group,in which participants will receive conventional integrated therapy on CRF.
- Integrated Therapy and colonic dialysis (Experimental): This arm is a treatment group,in which participants will receive integrated therapy on CRF and traditional Chinese medicine Colonic dialysis with traditional Chinese medicine colon lotion once a day.
  Interventions: Drug: colon lotion

INTERVENTIONS:
Drug: colon lotion — The colon lotion used in this clinic trial is a kind of hospital preparation. It is brown liquid,which consists of Rhubarb, Concha ostreae and some other traditional Chinese medicine.The colon lotion is diluted from 30ml to 150ml each time and will be used once a day for 10 days.
  Other Names: YZ20071408
  Arms: Integrated Therapy and colonic dialysis

SUMMARY:
This study evaluates the clinical efficacy and study the therapeutic mechanism of a kind of traditional Chinese medicine colonic dialysis on Chronic kidney disease (CKD) 5 without blood dialysis therapy in adults. Half of participants will receive conventional integrated therapy on chronic renal failure (CRF), while the other half will receive integrated therapy on CRF and traditional Chinese medicine colonic dialysis.

DETAILED DESCRIPTION:
Patients who would hospitalized in Nephrology of Guangdong Provincial Hospital of Traditional Chinese Medicine have chance to participate this study. All participates will be divided into two groups depending on their individual treatment interests and the baseline information will be balanced.

Integrated Therapy is routine symptomatic and supportive treatment for CRF,including reducing blood pressure and urine protein, improving anemia，regulating calcium and phosphorus metabolism and so on.The colon lotion used in colonic dialysis is a kind of hospital preparation. It consists of Rhubarb, Concha ostreae and some other traditional Chinese medicine.The whole treatment lasts about 10 days,as long as a regular drill-and-fill procedure. Before and after the treatment, related body dimensions will be tested.

ELIGIBILITY:
Inclusion Criteria:

* 1.corresponding to diagnosis standards of CKD-5:eGFR≤15ml/min/1.73m2; 2. did not receive kidney replacement therapy; 3. no gastrointestinal diseases (including ulcerative colitis, irritable bowel syndrome, inflammation, cancer, infection, bleeding, etc.) in the past 1 year; 4.not associated with rectal-related disorders (hemorrhoids, anal fistula, rectal cancer, cancer, infection, bleeding, etc.); 5.Sign informed consent.

Exclusion Criteria:

* 1. having used antibiotics, hormones, immunosuppressive, probiotics and laxatives in past three months; 2. pregnant or lactating patients; 3.cannot cooperate or tolerate colonic dialysis treatment; 4.combined with active stage of malignant tumors, cardiovascular, respiratory system, decompensated liver cirrhosis or blood system diseases (including coagulation disorders, hematopoietic dysfunction, etc.) and other serious primary disease; 5. recent merger of patients with infectious diseases; 6.having known to be allergic to some drugs in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-10-15 (Estimated)

PRIMARY OUTCOMES:
Change of glomerular filtration rate index | the first day before intervention and the eleventh day
  measuring the level of urea nitrogen，blood urea nitrogen,serum creatinine, serum cystatin C, blood and urineβ2-microglobulin. calculating the creatinine clearance rate.
Change of intestinal flora | the first day before intervention and the eleventh day
  measuring serum endotoxin and investigating the differences of intestinal flora between control group and experience group，as well as the differences between before colonic dialysis and after colonic dialysis.

SECONDARY OUTCOMES:
Change of serum electrolyte changes | the first day before intervention and the eleventh day
  measuring serum contents of sodium，potassium and phosphorus.
Change of related inflammatory index | the first day before intervention and the eleventh day
  measuring hs-C reactive protein(hs-CRP),interleukin 1β(IL-1β)，IL-6，tumor necrosis factor α(TNF-α) in serum.
Change of renal fibrosis index | the first day before intervention and the eleventh day
  measuring platelet derived growth factor (PDGF) secretion and serum transforming growth factor β(TGF-β).

CONTACTS AND LOCATIONS:
Overall Officials: Chen X Yin, Ph.D, Study Chair — Jinan University Guangzhou; Bao Kun, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine; Pang Peng, Principal Investigator — Jinan University Guangzhou
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Besides personal privacy information of the patients, all the other individual patient data（IPD）that treatment related will be shared with other researchers.After articles of this study publishing,researchers can obtain the information from the articles or sending e-mail to us.